CLINICAL TRIAL: NCT03680651
Title: Frequency and Type of Genetic Abnormalities Found in Antenatal Corpus Callosum Malformation
Acronym: AGMCC1318
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: AGMCC1318 (29BRC18.0123)
Record Dates: First submitted 2018-08-30; First posted 2018-09-21 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-06

CONDITIONS: Corpus Callosum Malformation; Prenatal Disorder
MeSH Terms: conditions — Agenesis of Corpus Callosum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Corpus callosum malformation (CCM) is the most frequently detected cerebral defect diagnosed in the prenatal setting. The most common CCM is corpus callosum agenesis (CCA) which is found in 2 to 3% of patients presenting with intellectual disability.

When CCM is diagnosed, the risk of chromosomal disorder is estimated to be 16%, be it aneuploidy such as trisomy 18, trisomy 13 or mosaic trisomy 8, or a chromosome structure anomaly, copy number variation or more complex rearrangement In France, since 2013 oligoarray-based comparative genomic hybridization (aCGH) analysis is performed in the prenatal period for most malformations after approval by a multidisciplinary prenatal diagnosis ethics committee (Centre Pluridisciplinaire de Diagnostic Prénatal, CPDPN) . However, to date only a few studies have been published which report recurrent Copy Number Variations (CNV) associated with CCM and estimate the risk for a chromosomal disorder, thus making counseling difficult in this context of prenatal diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Prenatal diagnosis of corpus callosum malformation, isolated or not, between 01/01/2013, and 31/05/2018
* Fetal DNA available
* Mother's informed consent obtained

Exclusion Criteria:

* No amniocentesis performed
* Refusing to participate

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Fetuses with prenatal diagnosis of corpus callosum malformation and antenatal molecular analysis by array CGH performed
Sampling Method: Non-Probability Sample
Enrollment: 275 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
frequency of chromosomal abnormalities | 6 months
  The main objective is to describe the frequency of chromosomal abnormalities associated with a prenatal diagnosis of corpus callosum agenesis in the hope of improving genetic counseling.

SECONDARY OUTCOMES:
Type of chromosomal abnormalities | 6 months
  Describe the type of chromosomal abnormalities associated with a prenatal diagnosis of corpus callosum agenesis and thus identify recurrent copy number variations.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France